CLINICAL TRIAL: NCT03710642
Title: Prazosin for Disruptive Agitation in Alzheimer's Disease (AD) (PEACE-AD)
Brief Title: Prazosin for Agitation in Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Collaborators: National Institute on Aging (NIA) (NIH); VA Puget Sound Health Care System (U.S. Federal Agency); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADC-042-PRAZ; 5U19AG010483 (NIH)
Record Dates: First submitted 2018-10-09; First posted 2018-10-18 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer's Disease; Disruptive Behavior
Keywords: Dementia; Agitation; PEACE-AD
MeSH Terms: conditions — Alzheimer Disease; Problem Behavior; Dementia; Psychomotor Agitation | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Prazosin) (Active Comparator): Eligible participants will be randomized using a 2:1 schedule to prazosin or placebo and stratified by site and gender, and will follow a fixed titration scheme for the first 15 days, followed by a flexible does titration from days 15-29, then a maintenance phase stable dose from days 29 to the end of the 12 weeks study period.
  Prazosin Fixed titration dose schedule for Days 1 to 14 1 mg QHS for Days 1 to 3
  1 mg QAM and 1 mg QHS for days 4 to 7
  1. mg QAM and 2 mg QHS for days 8 to 10
  2. mg QAM and 2 mg QHS for days 11 to 14
  Prazosin Flexible titration dose schedule for Days 15 to 29. 3 mg QAM and 3 mg QHS on day 15, 4 mg QAM and 4 mg QHS on day 22, 4 mg QAH and 6 mg QHS on day 29,
  Dose increases will be allowed only during the fixed and flexible dosing periods.
  Interventions: Drug: Prazosin
- Placebo oral capsule (Placebo Comparator): Placebo medication will be administered in a titration schedule mimicking the active comparator treatment.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Prazosin — Oral prazosin HCl capsules (or placebo) will be administered twice daily, with individualized doses up to a maximum of 4 mg QAM mid-morning and 6 mg at bedtime (QHS), or matching placebo capsules
  Other Names: Prazosin HCl; Minipress
  Arms: Treatment (Prazosin)
Drug: Placebo oral capsule — Placebo capsule matched to appearance of active drug.
  Other Names: Placebo
  Arms: Placebo oral capsule

SUMMARY:
The study evaluates the effects of Prazosin on agitation in adults with Alzheimer's disease.

Two thirds of the participants will participate in the medication portion, while one third will participate in the placebo portion

DETAILED DESCRIPTION:
Prazosin for Disruptive Agitation in Alzheimer's Disease (PEACE-AD) is a Phase IIb multicenter, randomized, double-blind, placebo-controlled trial of 12-weeks treatment with the brain active alpha-1 adrenoreceptor (AR) antagonist prazosin for disruptive agitation in 35 Alzheimer's disease (AD) residents in a long-term care (LTC) setting or living at home with full-time caregiving.

Distruptive agitation defined as having one or more of the following behaviors nearly daily during the previous week and at least intermittently for four weeks prior to screening: a) irritability, b) physically and/or verbally aggressive behavior, c) physically resistive to necessary care, d) and/or pressured motor activity (e.g., pressured pacing).

LTC is defined as assisted living or skilled nursing facility. Home dwelling participants require full-time caregiving defined as having continuous daily caregiving and a Study Partner who will assist in providing protocol specific information to the study team.

A previous single site pilot study addressing disruptive agitation in 22 predominantly LTC-residing AD participants demonstrated efficacy of prazosin on all three primary outcome measures.1 The current multicenter study is funded by the National Institute on Aging (NIA), and coordinated through the NIA-funded Alzheimer's Disease Cooperative Study (ADCS).

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria be included in the study:

1. Men and women with probable or possible AD by NINCDS-ADRDA criteria utilizing history; medical records review; physical and neurological exam; and laboratory tests (as applicable). Brain neuroimaging is not a requirement.
2. Participants must either reside in an LTC that is associated with the study site or at home with full-time caregiving.
3. Participants must have disruptive agitation significant enough to disrupt caregiving and, in the opinion of the Site Principal Investigator, to justify treatment. Disruptive agitation, defined as having any combination of the following target behaviors, must have occurred nearly daily during the previous week and at least intermittently for 4 weeks prior to screening:

   1. irritability,
   2. physically and/or verbally aggressive behavior,
   3. physical resistiveness to necessary care
   4. pressured motor activity (e.g., pressured pacing) These behaviors must be problematic in that they cause participant and caregiver distress and/or interfere with essential care or disrupt their living environment. Target behaviors may be any combination of the listed domains. Disruptive agitation must meet this threshold at Screening, documented on the Behavioral Inclusion Criteria Checklist.
4. Psychotropic medication, if used, should be stable for at least 2 weeks prior to randomization.
5. If taking cholinesterase inhibitor and/or memantine, must be on stable dose for 3 months prior t o randomization.
6. During the week before randomization, the above-described behaviors of eligible participants must be rated as of at least moderate severity.

Exclusion Criteria:

Participants meeting any of the following criteria must not be included in the study:

1. History of schizophrenia, schizoaffective disorder, or bipolar disorder according to the criteria of the most current version of the Diagnostic and Statistical Manual of Mental Disorders (DSM).
2. Other neurodegenerative diseases, including Parkinsons disease and Huntingtons disease, or cerebral tumor.
3. Dementia other than probable or possible AD per NINCDS-ADRDA criteria, such as human immunodeficiency virus (HIV) dementia, Creutzfeldt-Jakob disease, frontotemporal dementia, multiple cerebral infarctions, or normal pressure hydrocephalus.
4. Current treatment for seizure disorder (Note: anticonvulsants prescribed for disruptive agitation in the absence of seizure disorder will be allowed).
5. Abnormal laboratory values with clinical significance in the opinion of the site Principal Investigator.
6. Current unstable medical illness including delirium, worsening congestive heart failure, unstable angina, recent myocardial infarction (within the past 3 months), acute infectious disease, severe renal or hepatic failure, severe respiratory disease, metastatic cancer, or other conditions that, in the Site Principal Investigators opinion, could interfere with the analyses of safety and efficacy in this study.
7. Bedbound; participants may be ambulatory or use a wheelchair.
8. Absence of any comprehensible language.
9. Participation in another clinical trial for an investigational agent and took at least one dose of study drug (unless unblinded on placebo) within 12 weeks prior to screening. (The end of a previous investigational trial is defined as the date of the last dose of an investigational agent).
10. Preexisting recurrent hypotension (systolic BP <110).

    * If a reading of <110 systolic is measured at screening,
    * If the individual is taking antihypertensive medication: The Site PI should reassess the need for such medication and consider medication adjustments in consultation with the participants physician. One week following adjustment of antihypertensive(s), screening BP will be repeated for reassessment of eligibility. Further adjustment of antihypertensive medication regimen by the participants health care prescriber, may be indicated if systolic pressure remains <110. For inclusion, new systolic measurement following medication adjustment must be ≥110.
    * If the individual is not taking antihypertensive medication: repeat at least 3 BP measures over the course of 7-14 days. For inclusion, all three follow-up systolic measurements must be ≥110.
    * Any systolic reading <100 is exclusionary.
11. Preexisting orthostatic hypotension (>20 mmHg drop in systolic BP following 2 minutes of standing posture [or sitting if unable to stand] and accompanied by dizziness, lightheadedness, or syncope).
12. A 2-week washout is required prior to BL for the following exclusionary medications: prazosin or other alpha-1 blocker, sildenafil, vardenafil, tadalafil, and avanafil.
13. Women of childbearing potential are not included in this study. Women of non-childbearing potential are defined as any of the following:

    * have been postmenopausal (no menstrual cycle for past 24 months)
    * do not have a uterus,
    * have bilateral tubal ligation,
    * have undergone bilateral salpingectomy, and/or bilateral oophorectomy
14. The participant may not be an immediate family member of personnel directly affiliated with this study, the study site or funding agency. Immediate family is defined as a spouse, parent, child, or sibling, any of whom may be related by blood, adoption, or marriage.
15. P articipants whom the Site Principal Investigator deems to be otherwise unsuitable for participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Feldman, Principal Investigator — Alzheimer's Disease Cooperative Study (ADCS)
Locations (13):
- United States (13):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Southern California, Los Angeles, California
  - University of California, San Diego (UCSD), San Diego, California
  - Alta California Medical Group, Simi Valley, California
  - Stanford University, Stanford, California
  - University of Kentucky, Lexington, Kentucky
  - Northern Light/Acadia Hospital Eastern Maine Medical Center, Bangor, Maine
  - SUNY Upstate Medical University, Syracuse, New York
  - VAMC: James J Peters, The Bronx, New York
  - Oregon Health and Science University, Portland, Oregon
  - Roper St. Francis Hospital, Charleston, South Carolina
  - University of Texas, Health Science Center San Antonio, San Antonio, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data sharing is integral to the ADCS's mission to develop and execute innovative clinical trials focused on interventions that may prevent, delay, or treat the expression of Alzheimer's disease and related dementias. The ADCS is committed to sharing resources and tools, including data, biospecimens, trial designs, outcome and analysis measures following NIH guidelines.
  DATA SHARING: The ADCS Data and Sample Sharing Committee (DSSC) grants access to de-identified data to individuals who complete the request process and agree to the conditions in an ADCS/UCSD Data Use Agreement (DUA). After approval and receipt of the fully executed DUA, applicants are authorized to acquire data. Non-compliance with the DUA, including the requirement to provide requested updates will jeopardize further access to data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 01 March 2023
Access Criteria: Data requestors must complete an ADCS data and sample sharing request form. Upon approval, requestors must complete a data use agreement prior to accessing the data.
URL: https://www.adcs.org/data-sharing/

REFERENCES:
- [Background] Peskind ER, Wingerson D, Murray S, Pascualy M, Dobie DJ, Le Corre P, Le Verge R, Veith RC, Raskind MA. Effects of Alzheimer's disease and normal aging on cerebrospinal fluid norepinephrine responses to yohimbine and clonidine. Arch Gen Psychiatry. 1995 Sep;52(9):774-82. doi: 10.1001/archpsyc.1995.03950210068012. PMID 7654129
- [Background] Torroba Alvarez L, Hermida Donate JM, Ezpeleta Baquedano C, Munoz Zato E. [Methemoglobinemia secondary to the treatment of opportunistic infections in patients with AIDS]. Rev Clin Esp. 1988 Mar;182(5):289-90. No abstract available. Spanish. PMID 3399726
- [Background] Elrod R, Peskind ER, DiGiacomo L, Brodkin KI, Veith RC, Raskind MA. Effects of Alzheimer's disease severity on cerebrospinal fluid norepinephrine concentration. Am J Psychiatry. 1997 Jan;154(1):25-30. doi: 10.1176/ajp.154.1.25. PMID 8988954
- [Background] Raskind MA, Peskind ER, Holmes C, Goldstein DS. Patterns of cerebrospinal fluid catechols support increased central noradrenergic responsiveness in aging and Alzheimer's disease. Biol Psychiatry. 1999 Sep 15;46(6):756-65. doi: 10.1016/s0006-3223(99)00008-6. PMID 10494443
- [Background] Raskind MA, Peskind ER, Hoff DJ, Hart KL, Holmes HA, Warren D, Shofer J, O'Connell J, Taylor F, Gross C, Rohde K, McFall ME. A parallel group placebo controlled study of prazosin for trauma nightmares and sleep disturbance in combat veterans with post-traumatic stress disorder. Biol Psychiatry. 2007 Apr 15;61(8):928-34. doi: 10.1016/j.biopsych.2006.06.032. Epub 2006 Oct 25. PMID 17069768
- [Background] Raskind MA, Peterson K, Williams T, Hoff DJ, Hart K, Holmes H, Homas D, Hill J, Daniels C, Calohan J, Millard SP, Rohde K, O'Connell J, Pritzl D, Feiszli K, Petrie EC, Gross C, Mayer CL, Freed MC, Engel C, Peskind ER. A trial of prazosin for combat trauma PTSD with nightmares in active-duty soldiers returned from Iraq and Afghanistan. Am J Psychiatry. 2013 Sep;170(9):1003-10. doi: 10.1176/appi.ajp.2013.12081133. PMID 23846759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated September 2018: The research was initially approved for enrollment at Long Term Care facilities. Covid-19 impacted these facilities, and protocol amendments were approved to allow home-dwelling participants with full-time caregivers to enroll into the trial. Recruitment came from a blend of LTC facilities and institution/clinics.
Pre-assignment Details: Of the 54 participants consented and screened, 35 were eligible to participate in the trial and 19 were screening failures. Of the 35 participants randomized, 34 participants went on to receive study drug. One patient discontinued after randomization but prior to first dose administration.
Groups:
- Treatment (Prazosin): Eligible participants will be randomized using a 2:1 schedule to prazosin or placebo and stratified by site and gender, and will follow a fixed titration scheme for the first 15 days, followed by a flexible does titration from days 15-29, then a maintenance phase stable dose from days 29 to the end of the 12 weeks study period.
  Prazosin Fixed titration dose schedule for Days 1 to 14 1 mg QHS for Days 1 to 3
  1 mg QAM and 1 mg QHS for days 4 to 7
  1. mg QAM and 2 mg QHS for days 8 to 10
  2. mg QAM and 2 mg QHS for days 11 to 14
  Prazosin Flexible titration dose schedule for Days 15 to 29. 3 mg QAM and 3 mg QHS on day 15, 4 mg QAM and 4 mg QHS on day 22, 4 mg QAH and 6 mg QHS on day 29,
  Dose increases will be allowed only during the fixed and flexible dosing periods.
  Prazosin: Oral prazosin HCl capsules (or placebo) will be administered twice daily, with individualized doses up to a maximum of 4 mg QAM mid-morning and 6 mg at bedtime (QHS), or matching placebo capsules
Period: Overall Study
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Started | 27 | 8
Completed | 17 | 3
Not Completed | 10 | 5
Not completed — Adverse Event | 5 | 1
Not completed — non-site physician recommendation | 1 | 0
Not completed — Participant unwilling or unable to participate | 1 | 1
Not completed — "other" is selected as the reason for study termination | 1 | 3
Not completed — NA-no code provided | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants randomized to the clinical trial was a total of 35 participants. After randomization but before Investigational Product administration (IP= prazosin or placebo) one participant was withdrawn from the clinical trial, resulting in a total of 34 participants receiving IP. 26 participants received prazosin, 8 participants received placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule | Total
Number analyzed (Participants) | 26 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.02 (11.27) | 78.53 (8.0) | 79.67 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 6 | 25
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 21 | 8 | 29
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 8 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 8 | 34

OUTCOME MEASURES:

1. Primary Outcome: ADCS-Clinical Global Impression of Change in Agitation (ADCS-CGIC-A)
Description: The ADCS-CGIC-A is the primary outcome measure. It will be anchored to disruptive agitation, the target behaviors in this study. It measures whether the effects of active treatment are substantial enough to be detected by a skilled and experienced clinician on the basis of a direct examination of the participant and an interview of the participant's primary caregiver and other LTC facility staff. The baseline assessment is qualitative therefore there is no score at baseline; post-baseline scores represent a change score compared to baseline.
  The ADCS-CGIC-A is a 7-point scale that is structured as the clinician's assessment of change from baseline compared to the ADCS-CGIC-A Baseline Worksheet. There is no baseline score; post-baseline scores range from 1 (improvement) to 7 (worsening). A score of 1-2 indicates clinically meaningful improvement; a score of 3-5 indicates no clinically meaningful change; a score of 6-7 indicates clinically meaningful worsening.
Time Frame: From Baseline through Week 12.
Population: The population analyzed for this outcome includes: 20 study completers, and 3 early terminations that completed their termination visit at or after the week 10 timepoint. Therefore, the N analyzed is higher than the numbers of completers listed in the participant flow section.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 4
score on a scale | 3.434 (0.2833) | 3.442 (0.6141)
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.9904, Regression, Linear; Mean Difference (Net) = -0.008096

2. Secondary Outcome: Neuropsychiatric Inventory (NPI)/Neuropsychiatry Inventory-Nursing Home Version (NPI-NH)
Description: The NPI was designed to characterize the neuropsychiatric symptoms and psychopathology of patients with AD and other dementias residing in the community about which information was obtained from family caregivers. The content of the questions and their scoring in the NPI-NH are identical to those of the NPI except for some slight rephrasing to be consistent with the LTC environment where information is gathered from professional caregivers. Assessment of the impact of behavioral disturbances on family and professional caregivers, is assessed by a caregiver distress scale in the NPI and an occupational disruptiveness scale in the NPI-NH; scoring of this component remains identical. Minimum score is 0 and highest score is 144. A higher score means a worse outcome.
  This outcome is the change from baseline to week 12.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 24 | 7
units on a scale | -6.033 (4.692) | 5.506 (10.149)
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.30328, Regression, Linear; Mean Difference (Net) = -11.54

3. Secondary Outcome: Rescue Medication: Total mg Lorazepam Administered
Description: Cumulative total dose of Lorazepam rescue medication administered during the trial. Information on the total mg rescue lorazepam administered will be collected as additional secondary outcome measures. If prazosin is more effective than placebo, it is predicted that participants randomized to prazosin will be prescribed lower cumulative mg of rescue lorazepam for management of persistent or worsening disruptive agitation.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 24 | 7
mg | 0.25 (0.69) | 0.14 (0.24)
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.21981, Regression, Linear; Mean Difference (Net) = 0.31122

4. Secondary Outcome: Study Discontinuations
Description: Cox proportional hazard modelling comparing the median time to drop out between treatment groups.
Time Frame: 12 weeks
Measure: Median (Standard Deviation); unit: days
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 27 | 8
days | 65.63 (32.63) | 54.62 (33.29)
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.6366, Regression, Cox; Cox Proportional Hazard = -0.36277

5. Secondary Outcome: Responder Analysis on CGIC-A
Description: Comparison of proportions of responders versus non responders on the ADCS-CGIC-A. Responders are defined as those with moderate or marked improvement in agitation symptoms compared to baseline assessment.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 4
Participants | 7 | 1
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.9267, Regression, Logistic; Slope = -0.12842, Standard Error of Mean 1.39602

6. Secondary Outcome: ADCS-ADL-Severe
Description: The ADCS-ADL-Severe questionnaire is a secondary outcome measure aimed at detecting functional decline in people with severe AD. This scale is best suited for evaluating people with MMSE scores below 15/30, or equivalent. Questions are administered to a qualified caregiver informant about a set of 19 basic and instrumental ADL. Instrumental ADL are selected to be relevant to this level of severity of dementia, e.g., obtaining a beverage, turning lights on and off, turning a faucet on and off. Performance of each of these activities during the past 4 weeks, as well as the level of performance, are rated. A total score is derived by summing scores across items, and ranges from 0 (maximal impairment) to 54 (maximally independent function).
  This outcome is the change from baseline to week 12.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 4
score on a scale | -1.47055 (1.0062) | -4.53993 (2.1863)
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.2038, Regression, Linear; Mean Difference (Net) = 3.0694

7. Secondary Outcome: Caregiver Distress on NPI/NPI-NH
Description: Comparison of effects on caregiver distress/occupational disruptiveness scores on the NPI/NPI-NH. Minimum score is 0 and maximum score is 60. A higher score is a worse outcome.
  This outcome is the change from baseline to week 12.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
Number analyzed (Participants) | 19 | 4
score on a scale | -2.4438 (2.332) | 0.9446 (5.043)
Statistical Analysis 1: Comparison: Treatment (Prazosin) vs Placebo Oral Capsule; Test type: Superiority; p = 0.54133, Regression, Linear; Mean Difference (Net) = -3.388

8. Other Pre Specified Outcome: Cohen Mansfield Agitation Inventory (CMAI).
Description: The CMAI is an exploratory outcome measure for estimating frequency of agitated behaviors. The CMAI assesses the frequency of agitated behaviors in elderly persons and was developed for use in the LTC facility. The CMAI rates 29 agitated behaviors, each on a 7-point scale (1-7) of frequency ranging from never to several times per hour. Ratings pertain to the 2-week period preceding the rating. A higher score means a worse outcome.
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Five-domain NPI/NPI-NH Subset Score
Description: The Neuropsychiatric Inventory (NPI)/Neuropsychiatry Inventory-Nursing Home version (NPI-NH) subset score includes agitation/aggression, anxiety, disinhibition, irritability/lability and aberrant motor activity. Minimum and maximum values are 0 and 60 respectively. A higher score is a worse outcome.
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Sleep Continuity
Description: Actigraphy measures of locomotor activity during the night will be compared between groups.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from signed consent through the participant duration in the study. The specific time period is from consent through the end of the 12 week double-blind trial.
Arm/Group | Treatment (Prazosin) | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/8
Serious Adverse Events (participants affected / at risk) | 5/26 | 0/8
Other Adverse Events (participants affected / at risk) | 13/26 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Prazosin) (N=26) | Placebo Oral Capsule (N=8)
Syncope (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Prazosin) (N=26) | Placebo Oral Capsule (N=8)
Bradycardia (Cardiac disorders) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Syncope (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Anal incontinence (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 3 | 2
Lethargy (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 4 | 0
Pyrexia (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 1
Dizziness postural (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Somnolence (Psychiatric disorders) | 3 | 0
Incontinence (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Syncope (Vascular disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Following COVID-19, it became clear that it would not be possible to recruit the target sample size of 186 participants exclusively at LTC facilities. In 2021 we adjusted the trial size and incorporated the goal of gathering pilot data to demonstrate the feasibility of enrolling home dwelling participants and using remote visits. These changes resulted in the study sample size being re-estimated. Final enrollment was 35 randomized participants, of which 32 were at home with full time caregiving.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/42/NCT03710642/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT03710642/SAP_001.pdf
  • Informed Consent Form (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT03710642/ICF_002.pdf